CLINICAL TRIAL: NCT06998537
Title: The Effect of Spinal Anaesthesia on Haemodynamic Parameters in Patients Receiving Alpha Blockers
Brief Title: Hemodynamic Effects of Alpha Blockers in Patients With Spinal Anesthesia
Status: Not yet recruiting | Type: Observational
Sponsor: Izmir City Hospital (Other Government)
Responsible Party: Principal Investigator, Tuba Kuvvet Yoldaş, MD,Specialist, Izmir City Hospital
Other Study IDs: İSH-ANS-TK-01
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-07

CONDITIONS: Patient Group With Alpha Blocker Use
Keywords: spinal anesthesia; adrenergic α1-receptor antagonists,; Urologic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: α-1 adrenergic blocker users
- Group 2: No α-1 adrenergic blockers.

SUMMARY:
There is frequent use of alpha blockers in elderly patients with urological disorders. Various side effects are encountered due to the use of alpha blockers in the elderly age group. Especially hypotension is one of the common side effects. In addition, urological surgery is frequently performed in this age group. Spinal anesthesia is the most preferred anesthesia method in urological surgery. Spinal anesthesia may cause significant vasodilatation and thus hemodynamic changes such as hypotension by causing sympathetic nerve blockade. It is predicted that spinal anesthesia may increase these effects especially in individuals using α-1 adrenergic blockers. In the literature, serious hypotension has been encountered in individuals using alpha blockers under general anesthesia. The aim of this study was to compare the intraoperative hemodynamic changes in patients undergoing elective urologic surgery under spinal anesthesia between α-1 adrenergic blocker users (Group 1) and non-users(Group 2). Patients were divided into two groups according to drug use: Group 1: α-1 adrenergic blocker users (alfuzosin, doxazosin, terazosin,silodosin, tamsulosin), Group 2: No α-1 adrenergic blockers.

DETAILED DESCRIPTION:
Although α-1 adrenergic receptor blockers were initially developed for the treatment of hypertension, they have been widely used in the treatment of benign prostatic hyperplasia (BPH) over the last decade. α-1 adrenergic blockers are frequently used in the treatment of conditions such as benign prostatic hyperplasia (BPH) and lower urinary tract symptoms (LUTS), which are common in older age groups. α-1 adrenergic receptor blockers contribute to symptom relief by relaxing the smooth muscles of the prostate and bladder neck through inhibition of the sympathetic nervous system . However, blockers that are not receptor selective and cause vascular effects cause an increased risk of hypotension and dizziness when used at therapeutic levels. The hemodynamic effects of α-1 adrenergic blockers are a potential concern, especially in elderly patients. Physiologic changes with age, such as decreased cardiac output, impaired baroreceptor sensitivity, decreased plasma renin levels and renal function, make this patient group more vulnerable to complications related to vasodilation induced by α-blockers. This group of patients also frequently undergoes urological surgery and these procedures are usually performed under spinal anesthesia. Spinal anesthesia may cause significant vasodilatation and thus hemodynamic changes such as hypotension by causing sympathetic nerve blockade. It is predicted that these effects of spinal anesthesia may be increased especially in individuals using α-1 adrenergic blockers. However, there is insufficient data in the literature on the effect of α-1 adrenergic blocker use on intraoperative hemodynamic changes in patients undergoing spinal anesthesia. Existing publications have mostly focused on cases of severe hypotension after general anesthesia. The aim of this study was to compare the intraoperative hemodynamic changes in patients undergoing elective urologic surgery under spinal anesthesia between α-1 adrenergic blocker users(Group 1) and non-users(Group 2).

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists (ASA) physical status classification I,II or III over 18 years of age scheduled for elective urologic surgery under spinal anesthesia

Exclusion Criteria:

* Patients not undergoing spinal anesthesia, non-alpha-blocker vasoactive drug users, patients with cardiac disease, medical/surgical history of brain or spinal cord, neurological or psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective urologic surgery under spinal anesthesia
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Preop,15 minute,30minute mean arteriyal pressure | During procedure (From the beginning to the end of anesthesia)
  Hypotension MBP < 50 mmHg

SECONDARY OUTCOMES:
Preoperative, 15th and 30th minute heart rate | During procedure (From the beginning to the end of anesthesia)
  Bradycardia was defined as HR < 50 bpm

CONTACTS AND LOCATIONS:
Locations (1):
- İzmir City Hospital, Izmir, Bayraklı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No